CLINICAL TRIAL: NCT06477900
Title: Impact of SMS Reminder on Weight Loss, As Part of a Hygieno-dietary Health Pathway in Patients with Prediabetes: a Randomized Controlled Trial.
Brief Title: Impact of SMS Reminder on Weight Loss, As Part of a Health Pathway in Patients with Prediabetes (PREDIABCOACH)
Acronym: PREDIABCOACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/CHU/30
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMS receiption (Experimental): 150 participants will follow the FindRiscPei-CPTM program (current care) and will also receive 72 SMS messages over 6 months encouraging them to take part in sports and offering nutritional advice.
  Interventions: Other: SMS reception
- No SMS (No Intervention): 150 participants will only follow the FindRiscPei-CPTM program (current care) and will not receive SMS.

INTERVENTIONS:
Other: SMS reception — reception of 72 SMS encouraging physical activity and nutritional advice
  Arms: SMS receiption

SUMMARY:
The goal of this interventionnal study is to demonstrate that sending SMS messages with advice on physical activity or nutrition, in addition to a program of hygienic-dietary management, significantly increases weight loss in subjects with prediabetes in La Réunion.

Indeed, type 2 diabetes is a priority health problem on Reunion Island: 10% of the population are treated for type 2 diabetes, twice as many as in France.

International studies have demonstrated the value of modifying dietary and physical activity habits to reduce the risk of transition to diabetes in patients with prediabetes Against this backdrop, a Regional Nutrition Diabetes Program (PRND) 2020-2023 was launched by Réunion's Regional Health Agency (ARS) in 2020.

Studies have also demonstrated the effectiveness of using SMS to encourage and support weight loss interventions.

So, the main question it aims to answer are:

• Does the addition of 72 SMS of physical activity and nutriton advice, to the "FindRisc Péi-CPTS" program, significantly increase weight loss by 3% after 6 months of starting the program.

FindRiscPei-CPTS program includes sports sessions, dietary consultations and therapeutic education.

The 300 participants will be randomized into two arms

* 150 participants will take part in the FindRiscPei-CPTS program + receive SMS messages
* 150 participants will only take part in the FindRiscPei-CPTS program (no SMS)

All participants will follow procedures below:

* Inclusion: assessment of weight and waist circumference, Lifestyle Questionnaire and Socio-Efficacy Questionnaire.
* Participation in Findrisk program for 3 to 9 months (+ SMS for experimental group)
* 3 follow-up visits: 3 months, 6 months and 9 months after starting the program: weight and waist measurement, self-efficacy questionnaire.

DETAILED DESCRIPTION:
The outcomes of this study are :

* A better understanding of the effectiveness of the SMS intervention in the context of health and diet prevention programs for patients with pre-diabetes.
* More precise recommendations for healthcare professionals and decision-makers on the use of SMS intervention in this context.
* Improved health outcomes for prediabetes patients through the identification of effective diabetes prevention strategies.
* A positive impact on healthcare costs by reducing the progression from prediabetes to diabetes, and by reducing the use of costly healthcare associated with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subject with prediabetes as defined by HAS (fasting blood glucose > 1.10g/L and < 1.26g/L; or blood glucose 2h after ingestion of 10g of glucose > 1.40g/L and < 2g/L [HGPO test])
* included in a health and diet care program for patients with pre-diabetes offered by one of Réunion's CPTS (FindRisc Péi-CPTS program)
* age > 18 years
* in possession of an SMS-enabled telephone
* able to complete self-efficacy questionnaires
* not expected to move within 12 months

Exclusion Criteria:

* participant currently being monitored in the PREDIABRUN study
* protected adults (under guardianship or curatorship)
* pregnant women
* refusal to participate in the study
* patients unable to speak Creole or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Weight loss > 3% | 6 month
  Proportion of patients with weight loss greater than or equal to 3% at T1+6 months (comparison between FindRisc Pei-CPTS program + SMS intervention versus FindRisc Pei-CPTS program alone).

CONTACTS AND LOCATIONS:
Overall Officials: LERUSTE Sebastien, Dr, Principal Investigator — Réunion Island University
Locations (2):
- Communauté Professionnelle Territoriale de Santé (CPTS RéSO), Saint-Louis, Réunion, France
- Territorial Health Professional Community (CPTS) Grand Sud, Saint-Philippe, Reunion

IPD SHARING:
Plan to Share IPD: No